CLINICAL TRIAL: NCT05974085
Title: Prospective, Single-arm, Single-center, Phase II Clinical Study of XPO-1 Inhibitor Selinexor in Combination With RCHOP Regimen in the Treatment of Double Hit/Triple Hit B Cell Lymphoma
Brief Title: XPO-1 in Combination With RCHOP for DH/TH Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang haiyan, Director, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XRCHOP
Record Dates: First submitted 2022-01-13; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Double Hit Lymphoma; Triple Hit Lymphoma
Keywords: Double/Triple Hit Lymphoma; Selinexor; RCHOP

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selinexor+RCHOP (Experimental): Selinexor: 60 mg QW Rituximab: 375 mg/m2, d0 Vincristine: 4 mg, d1 Epirubicin: 75 mg/m2, d1 or Liposomal doxorubicin: 35 mg/m2, d1 Cyclophosphamide: 750 mg/m2, d1 Prednisone: 100 mg, d1-5
  Interventions: Drug: Selinexor+RCHOP

INTERVENTIONS:
Drug: Selinexor+RCHOP — XPO-1 inhibitor selinexor in combination with RCHOP

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of Selinexor in combination with RCHOP in first-line treatment of patients with DH or TH lymphoma.

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center clinical study evaluating the first-line treatment of DH or TH lymphoma with Selinexor combined with RCHOP. There are three stages: screening, treatment and follow-up period. The screening period was 28 days before the first dose. Treatment period: Enrolled subjects were treated with Selinexor in combination with RCHOP every 21 days for a maximum of 6 cycles until the efficacy of SD or PD, drug toxicity became intolerable, subject withdrawal of consent, death, or continuation of chemotherapy deemed unsuitable by the investigator. Lugano2014 criteria were used to evaluate the efficacy during treatment. Objective effective rate, safety and survival data were observed during the experiment. After stopping treatment or completing 6 cycles of treatment, subjects entered the follow-up period, during which imaging evaluation (enhanced CT at focal site is recommended) was performed at the following intervals: once every 3 months for 2 years, once every 6 months for 3-5 years, and once every 5 years until the end of the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical studies
2. Age: 18~75 (inclusive), male and female.
3. Histopathologically confirmed high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 gene rearrangement.
4. No previous chemotherapy, radiotherapy, immunotherapy or other anti-tumor therapy.
5. ECOG score is 0-2.
6. there must be at least one evaluable or measurable lesion that meets Lugano2014 criteria.
7. Adequate organ and bone marrow function.
8. Left ventricular ejection fraction (LVEF) ≥ 50% in cardiac function examination.
9. Serum pregnancy test negative

Exclusion Criteria:

1. Left ventricular ejection fraction (LVEF) ≥ 50% in cardiac function examination. 1) Mixed lymphoma (Hodgkin's lymphoma + non-Hodgkin's lymphoma), or DLBCL transformed from inert non-Hodgkin's lymphoma, or gray zone lymphoma (lymphoma between DLBCL and Hodgkin's lymphoma), or inert lymphoma with MYC, BCL2, BCL6 gene rearrangement.
2. known central nervous system involvement.
3. received prior anti-tumor therapy
4. Is participating in another clinical study or is receiving the first investigational drug less than 4 weeks after the completion of treatment in the previous clinical study
5. Had other malignant tumors in the past 5 years
6. Major surgery was performed within 28 days prior to study initiation
7. Cardiovascular function is unstable
8. Active infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From date of first day of treatment until the date of last day of treatment
  CR plus PR

SECONDARY OUTCOMES:
PFS | From date of first day of treatmentuntil the date of first documented progression, assessed up to 24 months
  Progression Free Survival
OS | From date of first day of treatmentuntil the date of first documented date of death from any cause, assessed up to 24 months
  Overall Survival
AE and SAE | From date of first day of treatmentuntil 30 day after last treatment
  Adverse event and serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Cong Li, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhenjiang, China

IPD SHARING:
Plan to Share IPD: No